CLINICAL TRIAL: NCT05900258
Title: Tirbanibulin 1% Ointment for the Treatment of Chronically Sun-damaged Skin on the Face
Acronym: SunDamage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunDamage
Record Dates: First submitted 2023-05-10; First posted 2023-06-12 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — tirbanibulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Tirbanibulin

INTERVENTIONS:
Drug: Tirbanibulin — Klisyri® 10 mg/g Ointment (Tirbanibulin) patients receive Tirbanibulin on sun-damaged areas of the face for five days, according to the SmPC.

SUMMARY:
Interventional, monocentric, national, single-arm, uncontrolled, open, prospective phase IV study. Since this study is not powered for confirmative testing, analysis is done by descriptive statistics Eligible AK patients receive Tirbanibulin on sun-damaged areas of the face for five days, according to the SmPC. Diagnosis and monitoring of treatment effects are supported by UV imaging using Canfield VISIA®. Safety and efficacy are assessed at end of treatment visit (EoT, approximately 3 days after the last dose, i.e, day 8 ± 2) and at a follow-up visit (FuV) 57 ± 7 d after the start of the treatment. UV images (Canfield VISIA®) will be taken at baseline, EoT and FuV, accompanied by conventional dermatological assessment according to clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosed with sun-damaged skin on the face and AK in the treatment area
* Willing and able to comply with all study procedures
* Use of medically acceptable contraception in males or females of child-bearing potential
* 51 -100 years of age
* Negative pregnancy test at baseline in females of childbearing potential

Exclusion Criteria:

* Allergy or intolerance towards the active ingredient or any of the constituents of the IMP
* Any contraindication for the IMP, according to the most recent version of the SmPC
* Open lesions of any kind on the face
* Concomitant cutaneous malignancy in treatment area, including but not restricted to squamous skin cancer
* Immune deficiency
* Participation in another clinical trial during the last six months
* Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Unmasking of subclinical lesions in UV-exposed areas of chronically sun-damaged skin of the face by a treatment with Tirbanibulin. | 57± 7 days
  Total clearance rates of unmasked lesions 57± 7 days after the start of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universität Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No